CLINICAL TRIAL: NCT01468051
Title: A Randomized Controlled Trial of Two Schedules of Hepatitis B Vaccination in Predialysis Chronic Renal Failure Patients
Brief Title: Two Schedules of Hepatitis B Vaccination in Predialysis Chronic Renal Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Khazaeipour, Principal Investigator, Nephrology Research Center, Department of Nephrology and Dialysis, Imam Khomeini Hospital., Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 507; 507 (Other: Tehran University of Medical Sciences)
Record Dates: First submitted 2011-10-27; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Renal Failure
Keywords: predialysed; chronic; renal failure patients
MeSH Terms: conditions — Renal Insufficiency; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 40 μg (2 ml) four doses of Euvax B vaccine (Experimental): 40 μg (2 ml) four doses of Euvax B vaccine (recombinant hepatitis B surface antigen adsorbed on aluminium hydroxide adjuvant- LG Chem, Korea)
  Interventions: Biological: four doses of Euvax B vaccine
- 20 μg (1 ml) three doses of Euvax B vaccine (Experimental): 20 μg (1 ml) three doses of Euvax B vaccine (recombinant hepatitis B surface antigen adsorbed on aluminium hydroxide adjuvant- LG Chem, Korea)
  Interventions: Biological: 20 μg (1 ml) three doses of Euvax B vaccine

INTERVENTIONS:
Biological: four doses of Euvax B vaccine — 40 μg (2 ml) four doses of Euvax B vaccine
  Other Names: Euvax B vaccine (recombinant hepatitis B surface antigen adsorbed on aluminium hydroxide adjuvant- LG Chem, Korea)
  Arms: 40 μg (2 ml) four doses of Euvax B vaccine
Biological: 20 μg (1 ml) three doses of Euvax B vaccine — 20 μg (1 ml) three doses of Euvax B vaccine (recombinant hepatitis B surface antigen adsorbed on aluminium hydroxide adjuvant- LG Chem, Korea)
  Arms: 20 μg (1 ml) three doses of Euvax B vaccine

SUMMARY:
Patients with chronic renal disease have to be vaccinated as soon as dialysis is forestalled and this could improve seroconversion rate of hepatitis B vaccination.

In this study, the investigators aimed to compare seroconversion rates and immune response rates using four doses of 40 μg and three doses of 20 μg of Euvax B recombinant hepatitis B surface antigen (HBsAg) vaccine given to predialysis CKD patients.

DETAILED DESCRIPTION:
In an open, randomized clinical trial, the investigators compared seroconversion rates in 51 predialysis patients with mild and moderate chronic renal failure using either 40 μg 4 doses or 20 μg 3 doses of Euvax B recombinant hepatitis B vaccine administered at 0, 1, 2, 6 and 0, 1, 6 months respectively.

ELIGIBILITY:
Inclusion Criteria:

* predialysis patients,
* > 18 years with mild and moderate chronic renal failure,
* serum creatinine between 1.5-6 mg/dl

Exclusion Criteria:

* patients with severe renal failure,
* serum creatinine > 6 mg/dl,
* requiring dialysis or expected to require dialysis within 1 year,
* receiving immunosuppressive treatment,
* known lymphoproliferative disorder.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Hepatitis B surface antibody mIU/ml | 8-10 weeks after the 6-month dose of vaccine
  Anti-HBs titres less than 10 mIU/ml were defined as non-seroconversion or non-responder. Anti-HBs titres greater than or equal to 10 mIU/ml but less than 100 mIU/ml were defined as seroconversion with low level antibody. Anti- HBs titres greater than or equal to100 mIU/ml were defined as seroconversion with protective levels of hepatitis B antibody.